CLINICAL TRIAL: NCT01047293
Title: A Phase I/II Study of RAD001, FOLFOX and Bevacizumab in Treatment of Colorectal Carcinoma
Brief Title: RAD001, FOLFOX and Bevacizumab in Treatment of Colorectal Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI38815
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Everolimus; Folfox protocol; Oxaliplatin; Fluorouracil; Leucovorin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All participants enrolled.
  Interventions: Drug: RAD001; Drug: FOLFOX; Drug: Bevacizumab

INTERVENTIONS:
Drug: RAD001 — RAD001 (everolimus) is a novel oral derivative of rapamycin.
  RAD001 is being investigated as an anticancer agent based on its potential to act:
  * Directly on the tumor cells by inhibiting tumor cell growth and proliferation
  * Indirectly by inhibiting angiogenesis leading to reduced tumor vascularity (via potent inhibition of tumor cell HIF-1 activity, VEGF production and VEGF-induced proliferation of endothelial cells). The role of angiogenesis in the maintenance of solid tumor growth is well established, and the mTOR pathway has been implicated in the regulation of tumor production of proangiogenic factors as well as modulation of VEGFR signaling in endothelial cells.
  Other Names: everlomius
Drug: FOLFOX — FOLFOX regimens combine oxaliplatin and leucovorin with bolus and infusional 5-fluorouracil (5-FU). 1 Oxaliplatin is a DNA cross-linking agent consisting of a platinum ion chelated with1, 2-diaminocyclohexane (DACH) and an oxalate ligand. It undergoes spontaneous activation in aqueous solutions via displacement of the labile oxalate ligand by water. The activated compounds bind with DNA, resulting in inter- and intra-strand platinum-DNA crosslinks. 5-FU is an anti-metabolite that blocks the methylation reaction of deoxyuridylic acid to thymidylic acid, causing thymidine-less cell death in rapidly growing cells. Leucovorin is reduced folic acid that modulates the activity of 5-FU by stabilizing the ternary 5-FdUMP/ thymidylate synthetase complex. Side effects associated with FOLFOX include neuropathy including pharyngo-laryngodysesthesia, diarrhea, nausea, vomiting, and mild myelosuppression.
  Other Names: oxaliplatin + 5 FU + leucovorin
Drug: Bevacizumab — Bevacizumab, a monoclonal antibody directed against VEGF (vascular endothelial growth factor) has been studied in a multitude of Phase I, II, and III clinical trials in more than 5000 patients in multiple tumor types. Phase III data in metastatic cancers
  Other Names: Avastin

SUMMARY:
RAD001 (everolimus) is a novel oral derivative of rapamycin. RAD001 has been in clinical development since 1996 as an immunosuppressant in solid organ transplantation and has obtained marketing authorization (Certican®) for prophylaxis of rejection in renal and cardiac transplantation in a number of countries, including the majority of the European Union. RAD001 has been in development for patients with various malignancies since 2002.

RAD001 is being investigated as an anticancer agent based on its potential to act:

* Directly on the tumor cells by inhibiting tumor cell growth and proliferation
* Indirectly by inhibiting angiogenesis leading to reduced tumor vascularity (via potent inhibition of tumor cell HIF-1 activity, VEGF production and VEGF-induced proliferation of endothelial cells). The role of angiogenesis in the maintenance of solid tumor growth is well established, and the mTOR pathway has been implicated in the regulation of tumor production of proangiogenic factors as well as modulation of VEGFR signaling in endothelial cells.

At weekly and daily schedules and at various doses explored, RAD001 is generally well tolerated. The most frequent adverse events (rash, mucositis, fatigue and headache) associated with RAD001 therapy are manageable. Non-infectious pneumonitis has been reported with mTOR inhibitors but is commonly low-grade and reversible.

Both FOLFOX and bevacizumab are well established for treatment of metastatic colorectal carcinomas. FOLFOX-6 can be combined safely with Bevacizumab and is currently in phase 3 testing for adjuvant therapy and is commonly used as a first line treatment regimen for metastatic colorectal cancers 25. There is an enhanced interest in development of more effective regimens for colorectal cancers. RAD001 is a mTOR inhibitor that has preclinical and clinical activity in colorectal cancers. RAD001 downregulates the mTOR pathway which can lead to direct antiproliferative effects as well as decreased production of Vascular Endothelial Growth Factor. A combination of RAD001 at 10 mg per day in combination with Bevacizumab 10 mg/kg every 2 weeks has been shown to be efficacious and safe. In another trial, RAD001 was shown to have many patients with stable disease and clearly needs to be given in combination therapy.

DETAILED DESCRIPTION:
Patient population Phase I portion: Metastatic colorectal cancer. A total of 3 patients on each cohort. Additional 3 patients on the tolerable cohort. Total patient number: Minimum 6, Maximum: 12 Phase II portion: Metastatic colorectal cancer: A total of 33 patients will be treated in this portion. This will include the patients treated on the tolerable dose level from the phase I trial. The statistical justification is indicated in the Statistics section 7.

Overall study design Phase I Study: A three cohort dose escalation will be used. Cycle length will be 28 days.

Bevacizumab FOLFOX-6 RAD001 Cohort 1: 5 mg/ kg Q 2weeks Standard Dose FOLFOX-6 2.5 mg PO qd Cohort 2: 5 mg/ kg Q 2weeks Standard Dose FOLFOX-6 5 mg PO qd Cohort 3: 5mg/kg Q 2 weeks Standard Dose FOLFOX-6 10 mg PO qd

Phase II Study:

For the Phase II portion the primary endpoint is Progression Free Survival at 6 months.

Study Objectives Primary

1. To evaluate the progression free survival (PFS) for a combination of FOLFOX+ Bevacizumab + RAD001 in previously untreated metastatic or advanced colorectal cancers
2. To evaluate the safety of the combination at a daily dosing of 2.5mg RAD001, 5 mg RAD001 or 10 mg RAD001 (Phase 1 part) Secondary

1. To study the toxicity profile of the combination 2. To study the Response Rate (RR) of the combination 3. To determine the serum proteomic profiles of patients treated with combination therapy (Both phase I and II portions)

Dose selection for RAD001 In phase 1 clinical studies of RAD001 as a monotherapy agent in oncology patients, the side-effect profile is essentially mild to moderate adverse events with a low frequency of DLT at the daily dose of 10 mg/d. Based on the PK/PD model, a daily dose of 10mg RAD001 is assumed to provide a persistently high degree of target inhibition in the tumor [Investigators' Brochure-Section 4.1.1.3]. In addition, preliminary data from phase 1 studies, in which changes in molecular characteristics of tumor induced by treatment with RAD001 at the doses of 5 and 10 mg/d were investigated, confirm the pharmacodynamic activity predicted previously by PK/PD modeling [Investigators' Brochure-Section 4.1.1.3]. Therefore, a dose of 10 mg/d should ensure adequate drug target inhibition for most patients, taking into consideration the known inter-patient variability in drug levels (CV of approx 50%). In this study, we will begin with a RAD001 dose of 2.5 mg which is the lowest dose that can be administered on a daily basis. If the dose is tolerable (<1/6 DLTs), we will escalate to the dose of RAD001 (5 mg) and a third cohort of 10 mg. If cohort 1 is intolerable, study will be closed without any further expansion. On any dose level, 3 patients would be enrolled. If there are 0/3 DLTs, we would be able to escalate the dose level. If 1/3 DLTs are observed, 3 additional patients will be enrolled on the same dose level. The intent is to escalate dose levels only if < 1/6 DLTs are observed. In case 2 or more DLTs are observed on a particular dose level, no further dose escalation is possible. This dose level would be deemed intolerable and the lower dose level would be expanded. The definition of the Maximum Tolerated Dose (MTD) is the highest dose level at which RAD001 can be combined with FOLFOX/ Bevacizumab with < 1/6 DLTs.

FOLFOX/ Bevacizumab: FOLFOX6 and Bevacizumab will be given as previously described 28. mFOLFOX6 (oxaliplatin 85 mg/m2 IV with LV 350 mg IV over 2 hours plus FU 400 mg/m2 IV bolus and 2,400 mg/m2continuous infusion over 46 hours every 2 weeks) will be combined with Bevacizumab given at 5 mg/kg every 2 weeks. Dose modifications will be carried out for chemotherapy as per the label for oxaliplatin, fluorouracil and bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced or metastatic colorectal cancers for whom chemotherapy is indicated
* Patients must not have had prior chemotherapy for advanced or metastatic disease. Patients could have received adjuvant chemotherapy or adjuvant chemo-radiotherapy
* Patients must have at least one measurable site of disease according to RECIST (version 1.1) criteria that has not been previously irradiated. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation
* Age ≥ 18 years
* Minimum of four weeks since any major surgery, completion of radiation, or completion of all prior systemic anticancer therapy (adequately recovered from the acute toxicities of any prior therapy)
* ECOG performance status £ 2
* Adequate bone marrow function as shown by: ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hgb > 9 g/dL
* Adequate liver function as shown by: serum bilirubin ≤ 1.5 x upper limit of normal (ULN), and serum AST and ALT ≤ 2.5 x ULN. With the exception of serum AST and ALT (< 5 x ULN) if the patient has liver metastases
* Adequate renal function, serum creatinine < 2 x ULN or creatinine clearance > 50 cc/hr
* Fasting serum cholesterol ≤300 mg/dL OR ≤ 7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In cases where one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication
* Signed informed consent
* INR and PTT < 1.5 (Anticoagulation is allowed if target INR < 1.5 on a stable dose of warfarin or on a stable dose of LMW heparin for > 2 weeks at time of randomization)

Exclusion Criteria:

* History of severe and uncontrolled allergic reactions to bevacizumab
* Symptomatic congestive heart failure of New York heart association Class III or IV
* Patients who have received prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus)
* DVT and hypertension controlled < 6 months
* Prior treatment with any investigational drug within the preceding 4 weeks
* Chronic treatment with systemic steroids or another immunosuppressive agent; topical or inhaled corticosteroids are allowed
* Patients should not receive immunization with attenuated live vaccines during study period or within 1 week of study entry
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Other malignancies that are active at the time of enrollment/ treatment on the protocol
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:
* unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤ 6 months prior to first study treatment, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
* severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air
* uncontrolled diabetes as defined by fasting serum glucose >1.5x ULN
* any active (acute or chronic) or uncontrolled infection/ disorders
* nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy
* known liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* A known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 in the judgment of the investigator (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis or on oral anti-vitamin K medication (except low dose Coumadin)
* Women who are pregnant or breast feeding, or women/men able to conceive and unwilling to practice an effective method of birth control. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of RAD001). Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study.
* Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Sharma, MD, Principal Investigator — Huntsman Cancer Institute
Locations (2):
- United States (2):
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Utah Cancer Specialists, Salt Lake City, Utah

REFERENCES:
- [Derived] Weldon Gilcrease G, Stenehjem DD, Wade ML, Weis J, McGregor K, Whisenant J, Boucher KM, Thorne K, Orgain N, Garrido-Laguna I, Sharma S. Phase I/II study of everolimus combined with mFOLFOX-6 and bevacizumab for first-line treatment of metastatic colorectal cancer. Invest New Drugs. 2019 Jun;37(3):482-489. doi: 10.1007/s10637-018-0645-2. Epub 2018 Oct 10. PMID 30302599

RESULTS

PARTICIPANT FLOW:
Groups:
- ARM 1 RAD001 5 mg QOD: Patients received 5mg RAD001 with FOLFOX and bevacizumab.
- ARM 2 5mg RAD001 QD: Patients received 5mg RAD001 QD with FOLFOX and bevacizumab.
- ARM 3 10mg RAD001 QD: Patients received 10mg RAD001 QD with FOLFOX and bevacizumab.
- ARM 4 10mg RAD001 QD - Phase II: Patients received 10 mg RAD001 with FOLFOX and bevacizumab. - Patient in the Dose Expansion Cohort not Dose Escalation
Period: Overall Study
Arm/Group | ARM 1 RAD001 5 mg QOD | ARM 2 5mg RAD001 QD | ARM 3 10mg RAD001 QD | ARM 4 10mg RAD001 QD - Phase II
Started | 4 | 8 | 9 | 26
Completed | 3 | 7 | 9 | 26
Not Completed | 1 | 1 | 0 | 0
Not completed — DLT criteria not fulfilled | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 47
Age, Continuous [Median (Full Range); unit: years] | 51 [23 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival at Six Months
Time Frame: 6 months
Population: Progression free survival at six month was calculated using all patients receiving one dose of drug therapy at all of the different dosing levels. The six month progression free survival was determined using Kaplan Meier methods
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 47
percentage of participants | 87 [76 to 99.9]

2. Primary Outcome: Evaluate Safety of the Combination at a Daily Dosing of 2.5mg RAD001, 5 mg RAD001 or 10 mg RAD001 (Phase 1 Part)
Description: Number of patients who experienced a Dose Limiting Toxicity (DLT). DLT will be assessed in the first 28 days of dosing. Patients need to get dosed with 2 rounds/sessions of all chemotherapy agents in the first 28 days in order to be evaluable for DLT assessment. The primary endpoint is safety as summarized by dose limiting toxicity (DLT).
Time Frame: December 2011
Measure: Number; unit: participants
Arm/Group | ARM 1 RAD001 5 mg QOD | ARM 2 5mg RAD001 QD | ARM 3 10mg RAD001 QD
Number analyzed (Participants) | 3 | 7 | 9
participants | 0 | 1 | 1

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 18/47
Other Adverse Events (participants affected / at risk) | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=47)
anemia (Blood and lymphatic system disorders) | 3 (4)
bowel perforation (Gastrointestinal disorders) | 4 (5)
c-diff infection (Infections and infestations) | 2 (3)
cholecystitis (Gastrointestinal disorders) | 1 (1)
confusion (Nervous system disorders) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 3 (3)
diarrhea (Gastrointestinal disorders) | 2 (2)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 2 (2)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
failure to thrive (Investigations) | 1 (1)
febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
fever (General disorders) | 2 (2)
fistula - small bowel (Gastrointestinal disorders) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infection - hepatic (Infections and infestations) | 1 (1)
Infection - pseudomonas (Infections and infestations) | 1 (1)
infection - urinary tract (Infections and infestations) | 2 (2)
Infections and other systemic inflammatory syndrome (Infections and infestations) | 1 (1)
left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
lipase increased (Metabolism and nutrition disorders) | 1 (1)
mucositis (Gastrointestinal disorders) | 4 (4)
muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 2 (3)
pain - abdominal (Gastrointestinal disorders) | 3 (3)
pain - chest (General disorders) | 1 (1)
pain - rectal/anal (Gastrointestinal disorders) | 1 (1)
pancreatitis (Gastrointestinal disorders) | 2 (2)
pericarditis (Cardiac disorders) | 1 (1)
pneumonia - aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary emboli (Vascular disorders) | 3 (3)
Renal calculi (Renal and urinary disorders) | 1 (1)
thrush (Infections and infestations) | 1 (1)
vasospasms (Vascular disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 1 (1)
weight loss (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=47)
body aches (General disorders) | 3 (4)
alkaline phosphatase increased (Metabolism and nutrition disorders) | 6 (7)
allergic reaction - anaphylactic (Immune system disorders) | 4 (5)
alopecia (Skin and subcutaneous tissue disorders) | 11 (12)
Alanine aminotransferase increased (Investigations) | 6 (8)
anemia (Blood and lymphatic system disorders) | 12 (22)
anorexia (Gastrointestinal disorders) | 25 (52)
anxiety (Psychiatric disorders) | 3 (4)
arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 5 (6)
ataxia (Nervous system disorders) | 3 (6)
bruising (Injury, poisoning and procedural complications) | 4 (4)
c-diff infection (Infections and infestations) | 3 (6)
confusion (Psychiatric disorders) | 3 (3)
congestion - sinus (Respiratory, thoracic and mediastinal disorders) | 13 (14)
constipation (Gastrointestinal disorders) | 12 (31)
cough (Respiratory, thoracic and mediastinal disorders) | 16 (28)
creatinine increased (Investigations) | 4 (6)
dehydration (Metabolism and nutrition disorders) | 20 (29)
depression (Psychiatric disorders) | 8 (10)
diarrhea (Gastrointestinal disorders) | 37 (86)
dizziness (Nervous system disorders) | 7 (7)
dry mouth (Gastrointestinal disorders) | 3 (3)
dry skin (Skin and subcutaneous tissue disorders) | 10 (12)
deep vein thrombosis (Vascular disorders) | 6 (6)
dysgeusia (Gastrointestinal disorders) | 18 (22)
dysphagia (Gastrointestinal disorders) | 8 (9)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (20)
dysuria (Renal and urinary disorders) | 3 (4)
edemia - penile/groin (General disorders) | 17 (25)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 29 (39)
fatigue (General disorders) | 43 (88)
fever (General disorders) | 12 (15)
flatulence (Gastrointestinal disorders) | 8 (8)
Erythroderma (Skin and subcutaneous tissue disorders) | 13 (23)
headache (Nervous system disorders) | 22 (27)
hematuria (Renal and urinary disorders) | 4 (5)
hemorrhage - rectal (Vascular disorders) | 3 (3)
hemorrhoids (Gastrointestinal disorders) | 5 (7)
hypercholesterolemia (Investigations) | 4 (5)
hyperglycemia (Metabolism and nutrition disorders) | 8 (13)
hypertension (Vascular disorders) | 12 (23)
hypertriglyceridemia (Metabolism and nutrition disorders) | 9 (15)
hypocalcemia (Metabolism and nutrition disorders) | 6 (7)
hypokalemia (Metabolism and nutrition disorders) | 17 (36)
hyponatremia (Metabolism and nutrition disorders) | 3 (4)
hypophosphatemia (Metabolism and nutrition disorders) | 12 (29)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (6)
infection - gums (Infections and infestations) | 3 (4)
infection - tooth (Infections and infestations) | 3 (3)
infection - urine/yeast (Infections and infestations) | 13 (29)
infection - vaginial (Infections and infestations) | 4 (8)
insomnia (Psychiatric disorders) | 10 (11)
leukopenia (Blood and lymphatic system disorders) | 16 (37)
lymphopenia (Blood and lymphatic system disorders) | 5 (7)
malaise (General disorders) | 3 (3)
mucositis (Gastrointestinal disorders) | 40 (146)
myalgia (Musculoskeletal and connective tissue disorders) | 7 (7)
nail changes (General disorders) | 7 (7)
nausea (Gastrointestinal disorders) | 37 (83)
neuropathy (Nervous system disorders) | 41 (95)
neutropenia (Blood and lymphatic system disorders) | 34 (102)
night sweats (General disorders) | 5 (5)
pain - unspecified (Gastrointestinal disorders) | 3 (3)
pain - abdominal (General disorders) | 21 (36)
pain - back (General disorders) | 14 (22)
pain - chest (General disorders) | 13 (17)
pain - extremity (General disorders) | 7 (11)
pain - rectal/anal (Gastrointestinal disorders) | 9 (16)
pain - shoulders (General disorders) | 3 (7)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (6)
post nasal drip (Respiratory, thoracic and mediastinal disorders) | 8 (8)
proteinuria (Renal and urinary disorders) | 8 (12)
pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 5 (5)
rash (Skin and subcutaneous tissue disorders) | 17 (25)
rash - acneiform (Skin and subcutaneous tissue disorders) | 3 (9)
rash - pruritic (Skin and subcutaneous tissue disorders) | 7 (8)
sore throat (Respiratory, thoracic and mediastinal disorders) | 14 (18)
tachycardia - sinus (Cardiac disorders) | 6 (8)
thrombocytopenia (Blood and lymphatic system disorders) | 16 (50)
thrush (Infections and infestations) | 9 (10)
toothache (General disorders) | 3 (3)
voice changes (General disorders) | 6 (7)
vomiting (Gastrointestinal disorders) | 25 (39)
weight loss (Investigations) | 28 (59)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes